CLINICAL TRIAL: NCT01029873
Title: Phase Ib/II Study of ALT-801 With Cisplatin in Patients With Metastatic Melanoma
Brief Title: QUILT-2.008: Study of ALT-801 With Cisplatin in Patients With Metastatic Melanoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Altor BioScience (Industry)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CA-ALT-801-02-09; R44CA097550 (NIH)
Record Dates: First submitted 2009-12-09; First posted 2009-12-10 (Estimated); Last update posted 2016-10-27 (Estimated); Status verified 2016-10

CONDITIONS: Metastatic Melanoma
Keywords: cancer; immunotherapy; targeted; metastatic; interleukin-2; IL-2; Cisplatin; antitumor; melanoma; TCR; T-cell receptor; p53; p53 gene; p53 tumor suppressor protein
MeSH Terms: conditions — Melanoma; Neoplasms; Neoplasm Metastasis | interventions — Cisplatin; ALT-801

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- ALT-801 (Experimental)
  Interventions: Drug: Cisplatin; Biological: ALT-801

INTERVENTIONS:
Drug: Cisplatin — Intravenous infusions; 2 treatment courses; 2 treatment cycles for each course; 70mg/m2 on day 1 of cycle 1 for each course
Biological: ALT-801 — Intravenous infusions; cycle 1: day 3 and 5; cycle 2: day 1, 3 and 5; nine day rest period between cycles; seven day recovery period between courses
  Stage 1: dose escalation (0.04 mg/kg, 0.06 mg/kg, 0.08 mg/kg)
  Stage 2: dose expansion (dose at MTD)

SUMMARY:
This is a Phase Ib/II, open-label, multi-center, competitive enrollment and dose-escalation study of ALT-801 combined with cisplatin. The purpose of this study is to evaluate the safety, determine the Maximum-Tolerated Dose (MTD), and characterize the pharmacokinetic profile of ALT-801 given with cisplatin in patients who are chemotherapy naïve and have metastatic melanoma that is considered surgically incurable. The anti-tumor responses of ALT-801 with cisplatin will also be assessed in this trial.

DETAILED DESCRIPTION:
Most current cancer treatment strategies involve the use of chemotherapeutic or biological drugs that exhibit variable efficacy and considerable toxicity. The limitations are often the result of the adverse side effects of the therapeutic drug on normal tissues. One approach to control these effects is to target the therapy to the tumor site. Of the identified tumor antigens, the human p53 tumor suppressor protein is overexpressed in a wide range of human malignancies. p53 is an intracellular tumor suppressor protein that acts to arrest the proliferation of cells. When mutated, it loses its ability to suppress abnormal proliferation and exhibits a longer half-life than the wild-type protein, allowing for its accumulation in tumors. In addition, p53 overexpression correlates with tumor transformation and aggression and is associated with lower overall survival rates and resistance to chemotherapeutic intervention in cancer patients. Therefore, p53 appears to be a marker for a considerable number of human malignancies and represents a good target for immunotherapeutics. However, p53 cannot be used as a target for antibodies because it is not displayed independently on the cell surface. Instead, the p53 protein is processed intracellularly into peptide fragments that are then displayed on the cell surface in the context of MHC. These peptide/MHC complexes are recognized by T-cells via their T-cell receptors (TCRs). Recently it has been confirmed that a p53 peptide fragment is significantly elevated in a wide range of human tumor tissues, particularly in melanoma, renal, lung, breast, colorectal, and osteosarcoma cancers. As a result, the feasibility of using soluble TCRs to target therapies against tumor cells that overexpress p53 is being investigated.

Interleukin-2 (IL-2) is a well-characterized growth factor for immune effector cells which play critical roles in tumor control and rejection. As a result, recombinant human IL-2 (e.g., Proleukin®, Chiron Novartis) has been approved for treatment of metastatic melanoma and renal cell carcinoma. IL-2 treatment provides significant benefit to a subset of patients with some maintaining durable responses for over ten years post-treatment. However, the major drawbacks of IL-2 therapy are its limited half-life and severe systemic toxicity. Hence, the use of high dose IL-2 is limited to specialized programs with experienced personnel, and it is generally offered to patients who are responsive and have excellent organ function. The low dose IL-2 treatment, while less toxic and more convenient, produces lower response rates and appears to be less effective in treating metastatic tumors. Thus, there is a critical need for innovative strategies that enhance the effects of IL-2 or reduce its toxicity without compromising clinical benefit. Targeted approaches to concentrate therapeutic cytokines, such as IL-2, at the tumor sites that express p53 could provide considerable advantages over current treatment.

The study drug, ALT-801, is a biologic compound composed of interleukin-2 (IL-2) genetically fused to a humanized soluble T-cell receptor directed against the p53-derived peptides expressed on tumor cells. This study is to evaluate whether directing IL-2 activity using ALT-801 to the patient's tumor sites that overexpress p53 results in clinical benefits if the ALT-801 treatment is given with cisplatin.

Platinum-based analogues including cisplatin, alone or in combination with other chemotherapies, have been shown to be active in patients with metastatic melanoma. Additionally, it is known that cisplatin, an alkylating agent known to inhibit DNA synthesis of dividing cells, triggers increased intracellular level of p53. The synergistic effects of cisplatin and ALT-801 treatment may induce cisplatin-mediated increases in p53 peptide display on the tumors and subsequently enhance tumor targeting of ALT-801.

ELIGIBILITY:
ENTRY CRITERIA:

DISEASE CHARACTERISTICS:

* Locally advanced or metastatic melanoma
* Measurable
* Histologically or cytologically confirmed
* Surgically incurable
* HLA-A2 positive and tumors that present HLA-A2.1/p53aa264-272 complexes

PRIOR/CONCURRENT THERAPY:

* If prior Proleukin treatment, must have had clinical benefit
* No prior systemic cytotoxic chemotherapy for melanoma
* No concurrent radiotherapy, chemotherapy, or other immunotherapy
* More than 4 weeks since prior major radiotherapy
* More than 8 weeks since prior CTLA-4 antagonist immunotherapy
* Not receiving other investigational agents

PATIENT CHARACTERISTICS:

Life expectancy

* > 3 months

Performance status

* ECOG 0 or 1

Bone marrow reserve

* Absolute neutrophil count (AGC/ANC) ≥ 1,500/uL
* Platelets ≥100,000/uL
* Hemoglobin ≥ 10g/dL

Renal function

* Serum creatinine ≤ 1.5 mg/dL

Hepatic function

* Total bilirubin ≤ 1.5 X ULN
* AST ≤ 2.5 X ULN
* Alkaline phosphatase ≤ 2.5 X ULN
* PT INR ≤ 1.5 X ULN
* aPTT ≤ 1.5 X ULN

Cardiovascular

* May be safely tapered off anti-hypertensives if currently on anti-hypertensives
* New York Heart Association classification I or II
* No congestive heart failure <6 months
* No unstable angina pectoris <6 months
* No myocardial infarction <6 months
* No history of ventricular arrhythmias
* Normal cardiac stress test required if any of the following is present:

  * Age ≥ 50
  * History of abnormal EKG
  * Symptoms of cardiac ischemia or arrhythmia

Pulmonary

* Normal pulmonary function test (FEV1 ≥ 70% of predicted value) if any of the following is present:

  * Prolonged history of cigarette smoking
  * Symptoms of respiratory dysfunction

Other

* No known autoimmune disease
* No known HIV positive
* No psychiatric illness/social situations that would limit study compliance
* No history or evidence of CNS disease
* No active systemic infection requiring parental antibiotic therapy
* No systemic steroid therapy required
* No prior organ allograft or allogeneic transplantation
* Not receiving chronic medication for asthma
* Not pregnant or nursing
* Fertile patients must use effective contraception

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2010-02; Primary Completion 2011-11 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety of the ALT-801-Cisplatin regimen. | 12 months
To assess the objective response (OR) which includes CR and PR. | 3 months
To assess the clinical benefit (CB) of the ALT-801-Cisplatin regimen which includes CR, PR and SD. | 3 months
To determine the MTD of the ALT-801-Cisplatin regimen. | 7 weeks

SECONDARY OUTCOMES:
To assess the six-month and one-year survival rates. | 12 months
To evaluate the immunogenicity and pharmacokinetic profile of ALT-801. | 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Hing Wong, PhD, Study Chair — Altor BioScience
Locations (8):
- United States (8):
  - The Angeles Clinic and Research Institute, Los Angeles, California
  - MD Anderson Cancer Center Orlando, Orlando, Florida
  - Emory University, Atlanta, Georgia
  - Northwestern University, Chicago, Illinois
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Carolinas Medical Center-Brumenthal Cancer Center, Charlotte, North Carolina
  - St. Luke's Hospital and Health Network, Bethlehem, Pennsylvania
  - University of Washington, Seattle Cancer Care Center, Seattle, Washington

REFERENCES:
- See also: Altor Bioscience Corporation, Miramar, Florida, US — http://www.altorbioscience.com